CLINICAL TRIAL: NCT06022887
Title: Feasibility and Acceptability of a Remote Time-Restricted Eating and Mindfulness-Based Stress Reduction Intervention to Reduce Risk Factors Associated With Early-Onset Colorectal Cancer Development Among Young Adults
Brief Title: Time-Restricted Eating and Mindfulness-Based Stress Reduction to Reduce the Risk of Early-Onset Colorectal Cancer
Acronym: MBSR&TRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lisa Tussing-Humphreys (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Sponsor-Investigator, Lisa Tussing-Humphreys, Professor, University of Illinois at Chicago
Organization: University of Illinois at Chicago (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY2023-0498
Record Dates: First submitted 2023-08-23; First posted 2023-09-05 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Obesity; Colorectal Cancer; Microbial Colonization; Time Restricted Feeding; Stress, Psychological
Keywords: obesity; Time Restricted Feeding; microbiome; chronic stress
MeSH Terms: conditions — Obesity; Colorectal Neoplasms; Communicable Diseases; Intermittent Fasting; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TRE alone (Experimental): Participants will be instructed to eat ad libitum from noon - 8:00pm daily and fast from 8:00pm - noon (16-h fast) for 8 weeks. During the 8-h eating window, there will be no restrictions on types or quantities of foods consumed. Participants will meet with a registered dietitian (RD) for 30 minutes at the start of the intervention to review instructions and goals and weekly thereafter. Adherence to the TRE intervention will be assessed as the number of adherent days per week.
  Interventions: Behavioral: TRE
- MBSR alone (Experimental): Participants in this study will be granted access to a remote mindfulness-based stress reductions (MBSR) protocol. Participants will have access to the MBSR course, consisting of 30 audio lessons, each ranging from 9 to 14 minutes long. During the study, participants will be asked to complete four lessons per week during weeks 1-7 and two lessons during week 8.
  Interventions: Behavioral: MBSR
- TRE + MBSR (Experimental): This group will follow a combined protocol of the TRE and MBSR interventions as described above.
  Interventions: Behavioral: TRE; Behavioral: MBSR
- Control (No Intervention): The control group will not receive any of the interventions previously described. To maintain a relationship with each participant in the control group, we will contact them once a week via text message to engage them to finalize the intervention period. At the end of the intervention period and after all data is collected, the RD will meet with the participant for 30 minutes and will educate them regarding the TRE protocol and provide access to the MBSR web-based program.

INTERVENTIONS:
Behavioral: TRE — daily ad libitum food intake, 8-h 12pm - 8pm, 8 wks active weight loss phase;
  Arms: TRE + MBSR; TRE alone
Behavioral: MBSR — Completed 30 sessions of a Mindfulness-Based Stress Reduction (MBSR) interventions for 8 weeks
  Arms: MBSR alone; TRE + MBSR

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility of remote time-restricted eating (TRE) and mindfulness-based stress reduction (MBSR) interventions and the preliminary effect on EOCRC-related markers. The main question[s] it aims to answer are:

* Is it feasible and acceptable to conduct 8-week remote interventions of TRE, MBSR, and combined TRE+MBSR among young adults with excess adiposity and moderate-to-severe perceived stress?
* Will participants in the combined group lose more body weight and reduce their stress levels than those in the remaining groups?
* Will participants in the combined group experience better body composition changes and improve their cardiometabolic health compared to those in the remaining groups?
* Will participants in the combined group exhibit changes in the microbiome compared to those in the remaining groups?

Participants will:

* Complete 8 weeks of a TRE intervention
* Complete 8 weeks of a remote MBSR intervention

Researchers will compare 1. TRE alone; 2. MBSR alone; 3. TRE + MBSR; and 4. Control to see if the study is feasible and acceptable; to see if individuals lose body weight; to see if individual stress levels reduce; to see changes in the microbiome.

DETAILED DESCRIPTION:
Early onset colorectal cancer (EOCRC) is defined as a diagnosis of colorectal cancer (CRC) in patients younger than 50 years old. The American Cancer Society reported that 12% of all CRC diagnoses as occurring in individuals younger than 50 years old. Worldwide, a steady increase in EOCRC cases is observed among Westernized countries, which suggests that similar risk factors and exposures within these developed countries are contributors to EOCRC. In particular, increased adiposity from an early age that persists through adulthood and chronic psychosocial stress are under investigation as drivers of the recent uptick in EOCRC in the United States (US) and other Westernized countries. Obesity in early adulthood is strongly associated with increased risk of EOCRC; in the US, obesity affects 42% of adults. In addition, obesity is associated with metabolic, hormonal, and immune perturbations that can promote gene mutations that drive EOCRC tumorigenesis. Chronic stress can negatively impact several different systems of the human body including the sympathetic nervous system (SNS)-related catecholamines, epinephrine and norepinephrine, and hypothalamic-pituitary-adrenal (HPA)-axis related hormones including adrenocorticotropic hormone and the glucocorticoid, cortisol. Due to the broad impact that exposure to chronic stress has in the human body, chronic stress has been linked to several diseases, including cancer. The gut and the brain are connected through a bidirectional system coined the gut-microbiota-brain axis (GMBA). Chronic stress can disrupt the SNS, HPA-axis and immune system, leading to a shift in gut microbial ecology and metabolic function that tips the balance to a more pro-inflammatory colonic state conducive to the formation of EOCRC. This study will examine if mitigating chronic stress and weight loss can modify EOCRC risk in young adults at risk of EOCRC. Accumulating evidence suggests that time-restricted eating (TRE), a type of intermittent fasting, produces a ~300-500 kcal/d energy deficit by limiting an individual's daily eating window to 4-8 hours each day. Mindfulness meditation is the practice of cultivating a moment-to-moment awareness of internal and external experience in an accepting and open manner. In 1990, Kabat-Zinn developed Mindfulness Based Stress Reduction (MBSR): an intervention with a goal of reducing stress, pain, and suffering. MBSR is associated with lower perceived stress and decreased circulating cortisol concentrations. Existing evidence suggests that MBSR also yields EOCRC preventive effects specific to body weight reduction, increase of insulin sensitivity and reduction of inflammation. We propose to conduct an 8-week 4-arm randomized-controlled study of 1. TRE alone; 2. MBSR alone; 3. TRE + MBSR; and 4. Control among 40 young adults with obesity (BMI ≥ 30 kg/m2) and moderate to severe perceived stress (Perceived Stress Score ≥14) to evaluate the feasibility of the interventions and preliminary effect on EOCRC-related markers. Data generated from this preliminary trial would serve in developing a fully powered efficacy trial testing TRE+MBSR for EOCRC prevention among young adults in the Chicagoland area.

ELIGIBILITY:
Inclusion Criteria:

1. 18-39 years old.
2. BMI 30-49.99 kg/m2.
3. Own and use a smartphone, computer, or tablet with access to the Internet.
4. Score ≥ 14 on the Perceived Stress Score (PSS) at screening.

Exclusion Criteria:

1. Have a personal or family history of EOCRC.
2. Have taken antibiotics in the previous 2 months.
3. Have an inflammatory bowel disease or genetic predisposition to EOCRC or CRC (e.g., Lynch syndrome);.
4. Any cancer diagnosis or cancer treatment in the past 12 months.
5. Consume >50 grams ethanol daily (approximately 4-5, 12 ounces beers).
6. Use combustible tobacco.
7. Have history of bariatric surgery or bowel resection.
8. Have an active infection.
9. Have type 1 or type 2 diabetes, immunodeficiency/autoimmune disorder, or inflammatory bowel disease.
10. Use fiber or pre-/probiotic supplements >3 days per week.
11. Currently taking corticosteroids medication - inhaled, topical, or oral in the past 2 months (affects cortisol measures).
12. Are on a weight-loss diet or involved in a formal weight-loss program or are not weight stable for 3 months (+/- 4.5 kg) prior to the study.
13. Females who are pregnant/trying to become pregnant.
14. Have schizophrenia (medication can affect study outcomes).
15. Have an eating window of <10 hours/day or are currently following an intermittent fasting pattern.
16. Night shift workers (shift passes midnight).
17. Present a history of eating disorder.
18. Currently taking weight loss medication.
19. Illegal drug use in the past month (not marijuana).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Feasibility of the study | Baseline; through study completion, an average of 9 weeks
  the number of people interested in the study, those who pass phone and in-person screenings, and those who decline enrollment and their reasons. Once enrolled, we will closely monitor attendance, data completeness, session attendance, asynchronous intervention usage, and loss to follow-up/withdrawal. To monitor participant progress, we will update the CONSORT participant flow diagram every week. Participants who withdraw voluntarily will be asked for their reasons.
Acceptability of the study | Week 4 of the intervention; through study completion, an average of 9 weeks
  Participants will complete the acceptability of intervention measure (scores range from 4-20 points with higher scores reflecting higher acceptability).

SECONDARY OUTCOMES:
Hair cortisol | Baseline; through study completion, an average of 9 weeks
  Objective stress markers will be measured via hair cortisol
Serum adrenocorticotropic hormone (ACTH) | Baseline; through study completion, an average of 9 weeks
  Objective stress markers will be measured via serum ACTH.
Serum cortisol | Baseline; through study completion, an average of 9 weeks
  Objective stress markers will be measured via serum cortisol.
Serum norepinephrine | Baseline; through study completion, an average of 9 weeks
  Objective stress markers will be measured via serum norepinephrine
Perceived Stress Scale. | Screening; through study completion, an average of 9 weeks
  The Perceived Stress Scale queries participants' perceptions of feeling stress during the last month. Responses were on a 5-point scale from "never" to "very often." Scores will be summed to indicate current stress levels, with higher scores suggesting greater perceived stress (≥ 14 indicates moderate to high perceived stress).
Body fat mass | Baseline; through study completion, an average of 9 weeks
  Body fat mass will be measured via whole body dual energy x-ray absorptiometry (DEXA) scan.
Body lean mass | Baseline; through study completion, an average of 9 weeks
  Body lean mass will be measured via whole body dual energy x-ray absorptiometry (DEXA) scan.
Body bone density | Baseline; through study completion, an average of 9 weeks
  Body bone density will be measured via whole body dual energy x-ray absorptiometry (DEXA) scan.
Triglycerides | Baseline; through study completion, an average of 9 weeks
  Will be measured from plasma by a commercial lab.
High sensitivity C-reactive protein. | Baseline; through study completion, an average of 9 weeks
  Will be measured from plasma by a commercial lab.
homeostasis model assessment-insulin resistance (HOMA-IR) | Baseline; through study completion, an average of 9 weeks
  calculated from fasting glucose and insulin using a standard formula.
Microbial Deoxyribonucleic acid (DNA) isolation: 16S on V4 region | Baseline; through study completion, an average of 9 weeks
  performed on stool using Microbial DNA isolation

CONTACTS AND LOCATIONS:
Overall Officials: Manoela Lima Oliveira, MS, RD, LDN, Principal Investigator — PhD Candidate; Lisa M Tussing-Humphreys, PHD, RD, Principal Investigator — Associate Professor, Kinesiology and Nutrition
Locations (1):
- Applied Health Sciences Building - University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sinicrope FA. Increasing Incidence of Early-Onset Colorectal Cancer. N Engl J Med. 2022 Apr 21;386(16):1547-1558. doi: 10.1056/NEJMra2200869. No abstract available. PMID 35443109
- [Background] Doubeni CA, Major JM, Laiyemo AO, Schootman M, Zauber AG, Hollenbeck AR, Sinha R, Allison J. Contribution of behavioral risk factors and obesity to socioeconomic differences in colorectal cancer incidence. J Natl Cancer Inst. 2012 Sep 19;104(18):1353-62. doi: 10.1093/jnci/djs346. Epub 2012 Sep 5. PMID 22952311
- See also: If you are interested in this research, please answer some eligibility questions in the survey linked here. — https://redcap.link/mbsrandtre